CLINICAL TRIAL: NCT06823193
Title: How Self-processing Affects Mental Time Travel: a Neuropsychological Study
Brief Title: The Impact of Self-processing on Mental Time Travel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Centro Studi e Ricerche in Neuroscienze Cognitive (Cesena) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ICS Maugeri CE 2717
Record Dates: First submitted 2025-01-27; First posted 2025-02-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Brain Injuries, Focal
Keywords: Mental Time Travel; Projection; Self/other distinction
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Healthy Participants; vmPFC patients; not-vmPFC patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy participants (Active Comparator): All participants performed the MTT task, the Age estimation task and the Lifeline task.
  Interventions: Behavioral: Mental Time Travel task; Behavioral: Age Estimation control task; Behavioral: Lifeline task
- vmPFC patients (Experimental): All participants performed the MTT task, the Age estimation task and the Lifeline task.
  Interventions: Behavioral: Mental Time Travel task; Behavioral: Age Estimation control task; Behavioral: Lifeline task
- not-vmPFC patients (Active Comparator): All participants performed the MTT task, the Age estimation task and the Lifeline task.
  Interventions: Behavioral: Mental Time Travel task; Behavioral: Age Estimation control task; Behavioral: Lifeline task

INTERVENTIONS:
Behavioral: Mental Time Travel task — A psychophysical task (D'Angelo et al., 2023) will be adopted. In this task, a projection in time will be "induced" by faces of different ages. Face stimuli will be presented with a short sentence describing a particular life event, commonly occurring around 60. Participants will perform a two-alternative forced-choice task under two experimental conditions. In the "past projection" condition, they will indicate whether it is "likely" or "unlikely" that the person of the face shown could have experienced the indicated event 10 years earlier. In the "future projection," they will indicate whether it is "likely" or "unlikely" that the person depicted will experience the indicated event in 10 years.
Behavioral: Age Estimation control task — In this task participants will estimate the age of the faces adopted as stimuli.
Behavioral: Lifeline task — In this task participants will be instructed to associated each event with the age at which they believe it typically occurred.

SUMMARY:
Mental time travel (MTT) refers to the ability to project oneself backward into the past or forward into the future to envision past and future events. This study examines the role of the ventromedial prefrontal cortex (vmPFC) in orienting toward past and future events during MTT.

DETAILED DESCRIPTION:
Mental Time Travel (MTT) is the ability to project oneself toward another specific temporal location, in the past or future subjective time. Specifically, it requires placing mental events on a subjective timeline by remembering the past or imagining the future. Regarding neural correlates, the subjective experience of remembering the past is associated with the lateral parietal cortex, especially in the inferior parietal lobule (IPL). The involvement of parietal areas in MTT for past events has been confirmed by neuropsychological and neuromodulation studies. Patients with neglect, following a lesion of the right parietal cortex, show a deficit in judging events that occurred before a specific temporal reference, suggesting an impairment in the representation of past events. Using transcranial alternate continuos stimulation (tACS) D'Angelo and colleagues (2023) showed that parietal beta frequencies selectively alter participants' ability to project into the past, but not into the future. Regarding future processing, the involvement of prefrontal cortex has been widely reported. The dorsolateral prefrontal cortex (dlPFC) plays a key role in planning, while the ventromedial prefrontal cortex (vmPFC) is involved in future scenario construction. In addition, vmPFC patients are unable to project into the future and anticipate events ahead, supporting a crucial role of the vmPFC in future construction.

Parietal and prefrontal areas are also involved in the processing of self-related information. In particular, the right lateral parietal cortex is more involved in retrieving self-related information than other-related information. Regarding the role of prefrontal regions in processing the self, the vmPFC shows greater activity when imagining a mental scenario related to the self rather than to another person.

To better understand MTT ability, two important questions arise from the review of the relevant literature. First, does self-related information affect our ability to mentally travel in time? If so, may these two processes interact in the same brain areas? VmPFC might be a good candidate for the interaction between future projection and self-processing: self-related stimuli could increase one's ability to "move" to future MTT.

Regarding past and self-related processing, the role of the right lateral parietal cortex is still unclear. IPL neural activity could underlie both processes, thus revealing a crucial centre for the interplay between MTT past projection and self-processing (autobiographical component of MTT).

The purpose of the present study is to investigate the influence of self-related stimuli in MTT tasks in patients with focal brain injury. Specifically, the authors will test for the first time whether the temporal distance between present time and the likelihood that a life event will occur (or has already occurred) is different whether the event is referred to one's own face or someone else's face.

ELIGIBILITY:
Inclusion Criteria:

* the absence of general cognitive impairment, assessed by neuropsychological testing
* the presence of a focal brain lesion will be adopted as an inclusion criterion for patients.

Exclusion Criteria:

* psychiatric disorders
* multiple brain lesions

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Likely Responses of events (Percentage) | At baseline
  If the vmPFC plays a crucial role in MTT, by activating and orienting to general knowledge about common life events, then vmPFC patients' probability judgments (% Likely Responses) in the MTT task should not be modulated coherently as a function of the perceived age of the portrayed faces and the Past vs. Future Projection condition.
  Considering the prominent role played by the vmPFC in future-oriented cognition, we expect that deficits in MTT would be more marked in the Future compared to the Past Projection condition.

SECONDARY OUTCOMES:
Temporal estimation of cultural prototypical life event (years) | At baseline
  The deficit found in MTT may be related to an impairment in activating general knowledge about common events. If this is the case, it should also result in an impairment in temporally placing cultural events appropriately on a time-line representing the duration of life (in years, from birth to death). Moreover, these difficulties in the temporal ordering of life events would be more marked for relatively future compared to relatively past events.

CONTACTS AND LOCATIONS:
Overall Officials: Giuliana Vezzadini, MD, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri, Castel Goffredo, Mantova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hutchinson JB, Uncapher MR, Wagner AD. Posterior parietal cortex and episodic retrieval: convergent and divergent effects of attention and memory. Learn Mem. 2009 May 23;16(6):343-56. doi: 10.1101/lm.919109. Print 2009 Jun. PMID 19470649
- [Background] Bonato M, Saj A, Vuilleumier P. Hemispatial Neglect Shows That "Before" Is "Left". Neural Plast. 2016;2016:2716036. doi: 10.1155/2016/2716036. Epub 2016 May 29. PMID 27313902
- [Background] Lou HC, Luber B, Crupain M, Keenan JP, Nowak M, Kjaer TW, Sackeim HA, Lisanby SH. Parietal cortex and representation of the mental Self. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6827-32. doi: 10.1073/pnas.0400049101. Epub 2004 Apr 19. PMID 15096584
- [Background] De Brigard F, Nathan Spreng R, Mitchell JP, Schacter DL. Neural activity associated with self, other, and object-based counterfactual thinking. Neuroimage. 2015 Apr 1;109:12-26. doi: 10.1016/j.neuroimage.2014.12.075. Epub 2015 Jan 8. PMID 25579447
- [Background] D'Argembeau A, Jedidi H, Balteau E, Bahri M, Phillips C, Salmon E. Valuing one's self: medial prefrontal involvement in epistemic and emotive investments in self-views. Cereb Cortex. 2012 Mar;22(3):659-67. doi: 10.1093/cercor/bhr144. Epub 2011 Jun 16. PMID 21680845
- [Background] Schacter DL, Addis DR, Hassabis D, Martin VC, Spreng RN, Szpunar KK. The future of memory: remembering, imagining, and the brain. Neuron. 2012 Nov 21;76(4):677-94. doi: 10.1016/j.neuron.2012.11.001. PMID 23177955
- [Background] Kaller CP, Rahm B, Spreer J, Weiller C, Unterrainer JM. Dissociable contributions of left and right dorsolateral prefrontal cortex in planning. Cereb Cortex. 2011 Feb;21(2):307-17. doi: 10.1093/cercor/bhq096. Epub 2010 Jun 3. PMID 20522540
- [Background] Ciaramelli E, Anelli F, Frassinetti F. An asymmetry in past and future mental time travel following vmPFC damage. Soc Cogn Affect Neurosci. 2021 Mar 5;16(3):315-325. doi: 10.1093/scan/nsaa163. PMID 33382070
- [Background] D'Argembeau A, Van der Linden M. Phenomenal characteristics associated with projecting oneself back into the past and forward into the future: influence of valence and temporal distance. Conscious Cogn. 2004 Dec;13(4):844-58. doi: 10.1016/j.concog.2004.07.007. PMID 15522635
- [Background] D'Angelo M, Frassinetti F, Cappelletti M. The Role of Beta Oscillations in Mental Time Travel. Psychol Sci. 2023 Apr;34(4):490-500. doi: 10.1177/09567976221147259. Epub 2023 Feb 16. PMID 37067986